CLINICAL TRIAL: NCT01274793
Title: Multicentre Randomized Controlled Trial for Quantity-Effect Relationship of Acupuncture With Two-ways Regulation to Treat Functional Enteropathy
Brief Title: Trial for Quantity-Effect Relationship of Acupuncture With Two-ways Regulation to Treat Functional Enteropathy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: The Fifth Hospital of Wuhan (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Guangying Huang, Institute of Integrated Traditional Chinese and Western Medicine, Tongji Hospital, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011CB505203
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Functional Constipation; Functional Diarrhea
Keywords: functional constipation; functional diarrhea; acupuncture
MeSH Terms: interventions — mosapride; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mosapride (Active Comparator): In the control group were orally administered 5 mg mosapride citrate tablet s three times a day for 4 continu ous weeks if no severe adverse effects were found.
  Interventions: Drug: Mosapride Citrate tablet
- Low-dose acupuncture (Experimental): In this low current intensity group, the current applied would be relatively weak,it was clearly perceived by the participants
  Interventions: Device: Low-dose acupuncture
- High-dose acupuncture (Experimental): In this group,the current was strong enough to reach the patients'tolerance threshold value.
  Interventions: Device: High-dose acupuncture

INTERVENTIONS:
Drug: Mosapride Citrate tablet — Orally administered 5 mg mosapride citrate tablet s three times a day for 4 continuous weeks if no severe adverse effects were found.
  Other Names: GASMOTIN
  Arms: Mosapride
Device: Low-dose acupuncture — In this low current intensity group, the current applied would be relatively weak,it was clearly perceived by the participants
  Arms: Low-dose acupuncture
Device: High-dose acupuncture — In this group,the current was strong enough to reach the patients'tolerance threshold value.
  Arms: High-dose acupuncture

SUMMARY:
the objective of this study is to investigate the Dose-Effect Relationship of Acupuncture with Two-ways Regulation Effect to Treat Functional Enteropathy

DETAILED DESCRIPTION:
eligibility criteria: functional constipation,functional diarrhea，irritable bowel syndrome

ELIGIBILITY:
Inclusion Criteria:

* function constipation function diarrhea

Exclusion Criteria:

* not function constipation not function diarrhea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2010-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
acupuncture benefits functional constipation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Guangying Huang, doctor, Study Director — institute of integrated traditional chinese and western medicine，Tongji meidical college,HUST
Locations (1):
- Institute of Integrated Traditional Chinese and Western Medicine, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Xu X, Zhang M, Wu X, Zheng C, Huang G. The Effect of Electroacupuncture Treatment with Different Intensities for Functional Diarrhea: A Randomized Controlled Trial. Evid Based Complement Alternat Med. 2022 Jan 4;2022:2564979. doi: 10.1155/2022/2564979. eCollection 2022. PMID 35027932
- [Derived] Zheng CH, Huang GY, Xu XH, Wang Y, Zhang MM, Wang W, Jing XH, Zhu B. Electro-acupuncture with different current intensities to treat functional constipation: a study protocol for a randomized controlled trial. Trials. 2013 Oct 22;14:344. doi: 10.1186/1745-6215-14-344. PMID 24143917